CLINICAL TRIAL: NCT00380744
Title: A Phase 1b/2 Multiple-Dose Safety Study and Pharmacokinetic/ Pharmacodynamic Study of LY2189102 in Patients With Rheumatoid Arthritis
Brief Title: A Safety and Pharmacokinetics Study in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8705; H9C-MC-BBDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2018-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — LY2189102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A LY2189102 0.1 mg/kg/wk (Experimental): Part A: 2 times (x) 0.1 milligrams/kilogram/week (mg/kg/wk) Loading dose, then 0.1 mg/kg/wk) X 4 weeks (wks), intravenous (IV)
  Part B: 2 x 0.02 mg/kg/wk Loading dose, then 0.02 mg/kg/wk X 4 wks, IV
  Interventions: Drug: LY2189102
- Part A LY2189102 0.3 mg/kg/wk (Experimental): Part A: 2 x 0.3 mg/kg/wk Loading dose, then 0.3 mg/kg/wk X 4 wks, IV
  Part B: 2 x 0.15 mg/kg/wk Loading dose, then 0.15 mg/kg/wk X 4 wks, IV
  Interventions: Drug: LY2189102
- Part A LY2189102 1.0 mg/kg/wk (Experimental): Part A: 2 x 1.0 mg/kg/wk Loading dose, then 1.0 mg/kg/wk X 4 wks, IV
  Part B: 2 x 1.0 mg/kg/wk Loading dose, then 1.0 mg/kg/wk X 4 wks, IV
  Interventions: Drug: LY2189102
- Part A LY2189102 2.5 mg/kg/wk (Experimental): Part A: 2 x 2.5 mg/kg/wk Loading dose, then 2.5 mg/kg/wk X 4 wks, IV
  Part B: 2 x 2.5 mg/kg/wk Loading dose, then 2.5 mg/kg/wk X 4 wks, IV
  Interventions: Drug: LY2189102
- Placebo (Placebo Comparator): IV, once weekly x 4 wks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LY2189102
  Arms: Part A LY2189102 0.1 mg/kg/wk; Part A LY2189102 0.3 mg/kg/wk; Part A LY2189102 1.0 mg/kg/wk; Part A LY2189102 2.5 mg/kg/wk
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of this antibody in participants with rheumatoid arthritis.

Part A of the study is an initial dose escalation phase

Part B of the study is a randomized allocation of the entire dosing group to parallel treatment assignments

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rheumatoid arthritis
* regular use of methotrexate
* active rheumatoid arthritis

Exclusion Criteria:

* Juvenile Rheumatoid Arthritis
* evidence of tuberculosis
* women who are pregnant or become pregnant during study, or are breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Orange, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayfield, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orangeburg, South Carolina
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw

REFERENCES:
- [Derived] Bihorel S, Fiedler-Kelly J, Ludwig E, Sloan-Lancaster J, Raddad E. Population pharmacokinetic modeling of LY2189102 after multiple intravenous and subcutaneous administrations. AAPS J. 2014 Sep;16(5):1009-17. doi: 10.1208/s12248-014-9623-6. Epub 2014 Jun 11. PMID 24912797
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow reports participants who discontinued from the study.
Groups:
- Part B - 0.02 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.04 milligrams/kilogram/week (mg/kg/wk) of LY2189102, followed by 0.02 mg/kg/wk for 4 weeks (wks), intravenously (IV).
- Part A - 0.1 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.2 mg/kg/wk of LY2189102, followed by 0.1 mg/kg/wk for 4 wks, IV.
- Part B - 0.15 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.3 mg/kg/wk of LY2189102, followed by 0.15 mg/kg/wk for 4 wks, IV.
- Part A - 0.3 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.6 mg/kg/wk of LY2189102, followed by 0.3 mg/kg/wk for 4 wks, IV.
- All Parts - 1.0 mg/kg/wk LY2189102: Participants were administered a loading dose of 2.0 mg/kg/wk of LY2189102, followed by 1.0 mg/kg/wk for 4 wks, IV.
- All Parts - 2.5 mg/kg/wk LY2189102: Participants were administered a loading dose of 5.0 mg/kg/wk of LY2189102, followed by 2.5 mg/kg/wk for 4 wks, IV.
- All Parts - Placebo: Participants were administered matched placebo IV, once weekly for 4 wks.
Period: Overall Study
Arm/Group | Part B - 0.02 mg/kg/wk LY2189102 | Part A - 0.1 mg/kg/wk LY2189102 | Part B - 0.15 mg/kg/wk LY2189102 | Part A - 0.3 mg/kg/wk LY2189102 | All Parts - 1.0 mg/kg/wk LY2189102 | All Parts - 2.5 mg/kg/wk LY2189102 | All Parts - Placebo
Started | 20 | 4 | 20 | 4 | 23 | 25 | 25
Received at Least 1 Dose of Study Drug | 20 | 4 | 20 | 4 | 23 | 25 | 25
Completed | 19 | 4 | 20 | 4 | 23 | 25 | 24
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Part B - 0.02 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.04 mg/kg/wk of LY2189102, followed by 0.02 mg/kg/wk for 4 wks, IV.
- Total: Total of all reporting groups
Arm/Group | Part B - 0.02 mg/kg/wk LY2189102 | Part A - 0.1 mg/kg/wk LY2189102 | Part B - 0.15 mg/kg/wk LY2189102 | Part A - 0.3 mg/kg/wk LY2189102 | All Parts - 1.0 mg/kg/wk LY2189102 | All Parts - 2.5 mg/kg/wk LY2189102 | All Parts - Placebo | Total
Number analyzed (Participants) | 20 | 4 | 20 | 4 | 23 | 25 | 25 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.1) | 52.5 (8.0) | 50.2 (14.7) | 51.7 (14.1) | 52.0 (12.4) | 54.0 (13.9) | 55.7 (10.6) | 53.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 2 | 17 | 4 | 16 | 15 | 22 | 93
  Male | 3 | 2 | 3 | 0 | 7 | 10 | 3 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 7
  Caucasian | 14 | 3 | 15 | 4 | 17 | 19 | 19 | 91
  Hispanic | 4 | 1 | 5 | 0 | 3 | 5 | 5 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 7 | 4 | 7 | 34
  Poland | 8 | 0 | 8 | 0 | 8 | 7 | 7 | 38
  Hungary | 3 | 0 | 3 | 0 | 3 | 3 | 3 | 15
  Argentina | 4 | 0 | 4 | 0 | 3 | 7 | 6 | 24
  Spain | 1 | 0 | 1 | 0 | 2 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs regardless of causality. A summary of s SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 98
Population: All data from all randomized participants who received at least 1 dose of study drug according to the assigned treatment.
  Per protocol analysis was performed per dose irrespective of study parts.
Measure: Count of Participants; unit: Participants
Groups:
- 0.02 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.04 mg/kg/wk of LY2189102, followed by 0.02 mg/kg/wk for 4 wks, IV.
- 0.1 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.2 mg/kg/wk of LY2189102, followed by 0.1 mg/kg/wk for 4 wks, IV.
- 0.15 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.3 mg/kg/wk of LY2189102, followed by 0.15 mg/kg/wk for 4 wks, IV.
- 0.3 mg/kg/wk LY2189102: Participants were administered a loading dose of 0.6 mg/kg/wk of LY2189102, followed by 0.3 mg/kg/wk for 4 wks, IV.
- 1.0 mg/kg/wk LY2189102: Participants were administered a loading dose of 2.0 mg/kg/wk of LY2189102, followed by 1.0 mg/kg/wk for 4 wks, IV.
- 2.5 mg/kg/wk LY2189102: Participants were administered a loading dose of 5.0 mg/kg/wk of LY2189102, followed by 2.5 mg/kg/wk for 4 wks, IV.
- Placebo: Participants were administered matched placebo IV, once weekly for 4 wks.
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Number analyzed (Participants) | 20 | 4 | 20 | 4 | 23 | 25 | 25
Participants
  SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Other Non-Serious AEs | 8 | 4 | 10 | 4 | 7 | 11 | 14

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve at Steady State for One Dosing Interval Time 0 to 168 Hours (AUC0-168 hr,ss) of LY2189102
Description: AUC0-168 hr,ss of individual participants was calculated by equation AUC=Dose/Clearance (CL), where the CL was estimated using a population PK model.
  Time frame for Part B: Day 1 predose, immediately after infusion (IAI), Day 14 and 28: predose and IAI, and Day 63 (Convenient time);
Time Frame: Part A: Day 1 predose and IAI, 2days post infusion, Day 14 and Day 28 predose and IAI, Day 35, 63 (convenient time)
Population: All participants who received at least 1 dose of study drug in part A & B and had evaluable AUC0-168 hr,ss results.
  Per protocol analysis was performed per dose irrespective of study parts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*h/mL)
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102
Number analyzed (Participants) | 20 | 4 | 20 | 4 | 23 | 25
micrograms*hour/milliliter (µg*h/mL) | 196 (52.5) | 902 (26.8) | 1150 (25.8) | 2810 (29.0) | 6650 (40.1) | 18200 (37.9)

3. Secondary Outcome: Change From Baseline in Simple Disease Activity Index Score (SDAI)
Description: SDAI is calculated as the sum of 5 components: tender joint count (TJC) and swollen joint count (SJC), Patient Global Assessment (PtGA) of disease activity visual analog scale (VAS) and Physician's Global Assessment of Disease Activity (PGA) VAS, and C-reactive protein (CRP). Total Score scale range is 0 (remission) to 86 (high disease activity). A negative change from baseline indicated an improvement. Least Squares (LS) mean calculated using a repeated measures model and adjusted for baseline + treatment + time + treatment * time.
Time Frame: Baseline, Days 7, 21, 35, 63, and 98
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 25 | 23
units on a scale
  Day 7: number analyzed (Participants) | 19 | 4 | 19 | 4 | 23 | 24 | 22
  Day 7 | -6.81 [-12.72 to -0.89] | -7.41 [-20.28 to 5.47] | -5.72 [-11.58 to 0.15] | -22.59 [-35.41 to -9.77] | -4.60 [-9.97 to 0.77] | -7.87 [-13.07 to -2.67] | -8.46 [-13.86 to -3.05]
  Day 21: number analyzed (Participants) | 20 | 4 | 18 | 4 | 23 | 25 | 21
  Day 21 | -13.96 [-19.80 to -8.12] | -19.61 [-32.48 to -6.74] | -10.78 [-16.74 to -4.83] | -26.16 [-38.98 to -13.34] | -14.85 [-20.22 to -9.48] | -13.57 [-18.71 to -8.42] | -11.70 [-17.18 to -6.22]
  Day 35 | -17.45 [-23.29 to -11.61] | -25.05 [-37.92 to -12.18] | -10.69 [-16.55 to -4.82] | -19.66 [-32.48 to -6.84] | -13.76 [-19.13 to -8.39] | -19.12 [-24.32 to -13.91] | -16.63 [-21.96 to -11.29]
  Day 63: number analyzed (Participants) | 20 | 4 | 19 | 4 | 21 | 25 | 23
  Day 63 | -17.73 [-23.57 to -11.89] | -20.48 [-33.36 to -7.61] | -9.27 [-15.14 to -3.41] | -21.72 [-34.54 to -8.90] | -14.14 [-19.64 to -8.63] | -19.49 [-24.63 to -14.35] | -13.02 [-18.36 to -7.68]
  Day 98: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 24 | 21
  Day 98 | -12.43 [-18.27 to -6.59] | -24.86 [-37.74 to -11.99] | -13.23 [-19.09 to -7.37] | -19.13 [-31.95 to -6.30] | -15.16 [-20.53 to -9.79] | -22.93 [-28.13 to -17.73] | -16.70 [-22.18 to -11.22]

4. Secondary Outcome: Change From Baseline in Disease Activity Score 28-Joint Count (DAS28)
Description: DAS28-4 (crp) is a modification of the original DAS based on TJC and SJC based on 28 joint counts, PGA VAS. DAS28-4 (crp) calculated as: 0.56*square root (sqrt) (TJC)+0.28*sqrt(SJC)+0.36*ln(CRP+1)+0.014*PGA+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity. A decrease in DAS28-CRP indicated an improvement in participant's condition.
  LS mean calculated using a repeated measures model and adjusted for baseline + treatment + time + treatment * time.
Time Frame: Baseline, Days 7, 21, 35, 63, and 98
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 25 | 23
units on a scale
  Day 7: number analyzed (Participants) | 19 | 4 | 19 | 4 | 23 | 24 | 22
  Day 7 | -0.71 [-1.18 to -0.25] | -0.68 [-1.69 to 0.33] | -0.50 [-0.96 to -0.05] | -1.66 [-2.66 to -0.65] | -0.48 [-0.91 to -0.06] | -0.59 [-0.99 to -0.18] | -0.61 [-1.04 to -0.19]
  Day 21: number analyzed (Participants) | 20 | 4 | 18 | 4 | 23 | 25 | 21
  Day 21 | -1.22 [-1.68 to -0.77] | -1.53 [-2.54 to -0.52] | -0.88 [-1.35 to -0.42] | -2.01 [-3.01 to -1.00] | -1.13 [-1.55 to -0.71] | -1.11 [-1.51 to -0.71] | -0.71 [-1.14 to -0.28]
  Day 35: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 24 | 23
  Day 35 | -1.43 [-1.89 to -0.98] | -1.99 [-3.00 to -0.99] | -0.84 [-1.29 to -0.38] | -1.43 [-2.44 to -0.43] | -1.06 [-1.48 to -0.64] | -1.56 [-1.96 to -1.15] | -1.04 [-1.46 to -0.62]
  Day 63: number analyzed (Participants) | 20 | 4 | 19 | 4 | 21 | 25 | 23
  Day 63 | -1.49 [-1.95 to -1.04] | -1.71 [-2.71 to -0.70] | -0.70 [-1.16 to -0.24] | -2.17 [-3.17 to -1.16] | -1.02 [-1.45 to -0.58] | -1.58 [-1.98 to -1.18] | -0.82 [-1.24 to -0.40]
  Day 98: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 24 | 21
  Day 98 | -1.06 [-1.51 to -0.60] | -2.25 [-3.25 to -1.24] | -1.08 [-1.54 to -0.63] | -1.84 [-2.84 to -0.83] | -1.23 [-1.65 to -0.81] | -1.89 [-2.29 to -1.48] | -1.11 [-1.54 to -0.68]

5. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is a biomarker associated with inflammation and structural damage. A negative change from baseline indicates improvement. LS mean calculated using a repeated measures model and adjusted for baseline + treatment + time + treatment * time.
Time Frame: Baseline, Days 7, 14, 21, 28, 35, 63, and 98
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams/deciliter (mg/dL)
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 25 | 24
milligrams/deciliter (mg/dL)
  Day 7: number analyzed (Participants) | 19 | 4 | 19 | 4 | 23 | 24 | 23
  Day 7 | -8.36 [-14.88 to -1.84] | -19.73 [-34.21 to -5.24] | -10.18 [-16.81 to -3.55] | -19.59 [-34.04 to -5.14] | -9.44 [-15.47 to -3.42] | -10.14 [-15.96 to -4.32] | -10.64 [-16.60 to -4.68]
  Day 14: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 25 | 23
  Day 14 | -9.43 [-15.89 to -2.97] | -19.86 [-34.35 to -5.38] | -8.33 [-14.96 to -1.70] | -21.02 [-35.47 to -6.57] | -10.88 [-16.90 to -4.85] | -8.29 [-14.07 to -2.51] | -9.04 [-15.00 to -3.07]
  Day 21: number analyzed (Participants) | 20 | 4 | 18 | 4 | 23 | 25 | 22
  Day 21 | -10.65 [-17.11 to -4.19] | -20.04 [-34.53 to -5.55] | -10.85 [-17.54 to -4.16] | -20.57 [-35.02 to -6.12] | -11.41 [-17.43 to -5.38] | -10.42 [-16.20 to -4.64] | -9.69 [-15.69 to -3.68]
  Day 28: number analyzed (Participants) | 20 | 4 | 19 | 4 | 22 | 25 | 23
  Day 28 | -12.43 [-18.90 to -5.97] | -19.61 [-34.10 to -5.13] | -9.63 [-16.26 to -3.00] | -20.76 [-35.21 to -6.31] | -13.53 [-19.60 to -7.46] | -10.27 [-16.05 to -4.49] | -12.05 [-18.02 to -6.09]
  Day 35: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 24 | 24
  Day 35 | -11.06 [-17.52 to -4.59] | -19.18 [-33.67 to -4.70] | -11.51 [-18.14 to -4.88] | -19.60 [-34.05 to -5.15] | -12.10 [-18.13 to -6.08] | -13.66 [-19.48 to -7.83] | -11.60 [-17.53 to -5.68]
  Day 63: number analyzed (Participants) | 20 | 4 | 19 | 4 | 21 | 25 | 24
  Day 63 | -11.26 [-17.72 to -4.79] | -19.01 [-33.50 to -4.52] | -10.23 [-16.86 to -3.60] | -20.69 [-35.14 to -6.24] | -10.29 [-16.41 to -4.17] | -8.66 [-14.44 to -2.88] | -9.05 [-14.98 to -3.13]
  Day 98: number analyzed (Participants) | 20 | 4 | 19 | 4 | 23 | 24 | 22
  Day 98 | -7.37 [-13.83 to -0.91] | -19.30 [-33.79 to -4.81] | -12.94 [-19.57 to -6.31] | -20.73 [-35.18 to -6.28] | -13.68 [-19.70 to -7.65] | -13.35 [-19.17 to -7.53] | -8.90 [-14.91 to -2.89]

6. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score
Description: HAQ was a participant-reported questionnaire that consisted of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do). The highest score for any question in a category was the score of that category unless special aids or devices or help from another person was required. Answers for at least 6 of the 8 disability domains were required to compute the participant's HAQ score. If the participant had scores for fewer than 6 categories, the HAQ score was considered missing. The HAQ score was calculated as the sum of the category scores divided by the number of categories scored, with a possible scores range from 0 to 3. Negative mean changes from baseline indicated improvement.
Time Frame: Baseline, Days 35, 63, and 98
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Number analyzed (Participants) | 20 | 4 | 20 | 4 | 23 | 25 | 24
units on a scale
  Day 35 | -0.22 [-0.44 to -0.00] | -0.09 [-0.58 to 0.40] | -0.09 [-0.30 to 0.13] | -0.22 [-0.71 to 0.26] | -0.19 [-0.39 to 0.02] | -0.71 [-0.90 to -0.51] | -0.29 [-0.49 to -0.09]
  Day 63 | -0.22 [-0.44 to -0.00] | -0.15 [-0.64 to 0.34] | -0.04 [-0.25 to 0.18] | -0.04 [-0.52 to 0.45] | -0.19 [-0.39 to 0.01] | -0.72 [-0.91 to -0.52] | -0.28 [-0.48 to -0.08]
  Day 98 | -0.25 [-0.46 to -0.03] | -0.34 [-0.83 to 0.15] | -0.11 [-0.32 to 0.11] | -0.13 [-0.62 to 0.36] | -0.18 [-0.38 to 0.03] | -0.75 [-0.95 to -0.56] | -0.31 [-0.51 to -0.11]

ADVERSE EVENTS:
Arm/Group | 0.02 mg/kg/wk LY2189102 | 0.1 mg/kg/wk LY2189102 | 0.15 mg/kg/wk LY2189102 | 0.3 mg/kg/wk LY2189102 | 1.0 mg/kg/wk LY2189102 | 2.5 mg/kg/wk LY2189102 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/4 | 0/20 | 0/4 | 0/23 | 1/25 | 2/25
Other Adverse Events (participants affected / at risk) | 8/20 | 4/4 | 10/20 | 4/4 | 7/23 | 11/25 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.02 mg/kg/wk LY2189102 (N=20) | 0.1 mg/kg/wk LY2189102 (N=4) | 0.15 mg/kg/wk LY2189102 (N=20) | 0.3 mg/kg/wk LY2189102 (N=4) | 1.0 mg/kg/wk LY2189102 (N=23) | 2.5 mg/kg/wk LY2189102 (N=25) | Placebo (N=25)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 0.02 mg/kg/wk LY2189102 (N=20) | 0.1 mg/kg/wk LY2189102 (N=4) | 0.15 mg/kg/wk LY2189102 (N=20) | 0.3 mg/kg/wk LY2189102 (N=4) | 1.0 mg/kg/wk LY2189102 (N=23) | 2.5 mg/kg/wk LY2189102 (N=25) | Placebo (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 3 (3) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0/17 (0) | 0/2 (0) | 1/17 (1) | 0 (0) | 0/16 (0) | 0/15 (0) | 0/22 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days